CLINICAL TRIAL: NCT03169959
Title: A Randomised, 3-Period, 3-Treatment, Single-dose, Open-label, Single-center, Crossover Study to Assess the Fed-state Bioequivalence of a Triple Fixed-Combination Drug Product of 2.5 mg Saxagliptin / 5 mg Dapagliflozin / 1000 mg Metformin XR and 5 mg Saxagliptin / 10 mg Dapagliflozin / 1000 mg Metformin XR Relative to Individual Components (Onglyza® and XIGDUO® XR) Co-administered to Healthy Subjects
Brief Title: A Study to Evaluate the Food Effect on Drug Availability, Pharmacokinetic (PK) Properties, Safety and Tolerability of Two Different Dose Combination Therapy of Saxagliptin/Dapagliflozin/Metformin Extended-release (XR) Against Individual Component Co-administration.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D168AC00001
Record Dates: First submitted 2017-05-23; First posted 2017-05-30 (Actual); Last update posted 2017-08-14 (Actual); Status verified 2017-08

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Anti-diabetic; Anti-hyperglycemic agents; Bioequivalence; Fixed-Combination Drug Product (FCDP) of saxagliptin / dapagliflozin / metformin extended-release (XR).; Fed-state bioequivalence (BE); XIGDUO® XR; ONGLYZA®
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — saxagliptin; dapagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- Cohort 1: Sequence 1 (ABC) (Experimental): Subjects were randomized to treatment sequence 1 ABC:
  On Day 1, each subjects will receive orally single-dose of the treatment assigned to that treatment period.
  A= Reference product - 2.5mg ONGLYZA (2.5mg saxagliptin) and 5/1000mg XIGDUO XR (5 mg dapagliflozin / 1000mg Metformin XR) after food.
  B = Test product - Triple FCDP consisting of 2.5 mg saxagliptin / 5 mg dapagliflozin / 1000 mg metformin XR after food.
  C = Test product - Triple FCDP tablet consisting of 2.5 mg saxagliptin / 5 mg dapagliflozin / 1000 mg metformin XR without food.
  Interventions: Drug: 2.5 mg Saxagliptin tablet; Drug: 5 mg dapagliflozin / 1000 mg metformin XR tablet; Drug: Triple FCDP - 2.5 mg saxagliptin / 5 mg dapagliflozin / 1000 mg metformin XR
- Cohort 1: Sequence 2 (ACB) (Experimental): Subjects were randomized to treatment sequence 1 ACB:
  On Day 1, each subjects will receive orally single-dose of the treatment assigned to that treatment period.
  A= Reference product - 2.5mg ONGLYZA (2.5mg saxagliptin) and 5/1000mg XIGDUO XR (5 mg dapagliflozin / 1000mg Metformin XR) after food.
  B = Test product - Triple FCDP consisting of 2.5 mg saxagliptin / 5 mg dapagliflozin / 1000 mg metformin XR after food.
  C = Test product - Triple FCDP tablet consisting of 2.5 mg saxagliptin / 5 mg dapagliflozin / 1000 mg metformin XR without food.
  Interventions: Drug: 2.5 mg Saxagliptin tablet; Drug: 5 mg dapagliflozin / 1000 mg metformin XR tablet; Drug: Triple FCDP - 2.5 mg saxagliptin / 5 mg dapagliflozin / 1000 mg metformin XR
- Cohort 1: Sequence 3 (BAC) (Experimental): Subjects were randomized to treatment sequence 1 ABC:
  On Day 1, each subjects will receive orally single-dose of the treatment assigned to that treatment period.
  A= Reference product - 2.5mg ONGLYZA (2.5mg saxagliptin) and 5/1000mg XIGDUO XR (5 mg dapagliflozin / 1000mg Metformin XR) after food.
  B = Test product - Triple FCDP consisting of 2.5 mg saxagliptin / 5 mg dapagliflozin / 1000 mg metformin XR after food.
  C = Test product - Triple FCDP tablet consisting of 2.5 mg saxagliptin / 5 mg dapagliflozin / 1000 mg metformin XR without food.
  Interventions: Drug: 2.5 mg Saxagliptin tablet; Drug: 5 mg dapagliflozin / 1000 mg metformin XR tablet; Drug: Triple FCDP - 2.5 mg saxagliptin / 5 mg dapagliflozin / 1000 mg metformin XR
- Cohort 1: Sequence 4 (BCA) (Experimental): Subjects were randomized to treatment sequence 1 ABC:
  On Day 1, each subjects will receive orally single-dose of the treatment assigned to that treatment period.
  A= Reference product - 2.5mg ONGLYZA (2.5mg saxagliptin) and 5/1000mg XIGDUO XR (5 mg dapagliflozin / 1000mg Metformin XR) after food.
  B = Test product - Triple FCDP consisting of 2.5 mg saxagliptin / 5 mg dapagliflozin / 1000 mg metformin XR after food.
  C = Test product - Triple FCDP tablet consisting of 2.5 mg saxagliptin / 5 mg dapagliflozin / 1000 mg metformin XR without food.
  Interventions: Drug: 2.5 mg Saxagliptin tablet; Drug: 5 mg dapagliflozin / 1000 mg metformin XR tablet; Drug: Triple FCDP - 2.5 mg saxagliptin / 5 mg dapagliflozin / 1000 mg metformin XR
- Cohort 1: Sequence 5 (CAB) (Experimental): Subjects were randomized to treatment sequence 1 ABC:
  On Day 1, each subjects will receive orally single-dose of the treatment assigned to that treatment period.
  A= Reference product - 2.5mg ONGLYZA (2.5mg saxagliptin) and 5/1000mg XIGDUO XR (5 mg dapagliflozin / 1000mg Metformin XR) after food.
  B = Test product - Triple FCDP consisting of 2.5 mg saxagliptin / 5 mg dapagliflozin / 1000 mg metformin XR after food.
  C = Test product - Triple FCDP tablet consisting of 2.5 mg saxagliptin / 5 mg dapagliflozin / 1000 mg metformin XR without food.
  Interventions: Drug: 2.5 mg Saxagliptin tablet; Drug: 5 mg dapagliflozin / 1000 mg metformin XR tablet; Drug: Triple FCDP - 2.5 mg saxagliptin / 5 mg dapagliflozin / 1000 mg metformin XR
- Cohort 1: Sequence 6 (CBA) (Experimental): Subjects were randomized to treatment sequence 1 ABC:
  On Day 1, each subjects will receive orally single-dose of the treatment assigned to that treatment period.
  A= Reference product - 2.5mg ONGLYZA (2.5mg saxagliptin) and 5/1000mg XIGDUO XR (5 mg dapagliflozin / 1000mg Metformin XR) after food.
  B = Test product - Triple FCDP consisting of 2.5 mg saxagliptin / 5 mg dapagliflozin / 1000 mg metformin XR after food.
  C = Test product - Triple FCDP tablet consisting of 2.5mg saxagliptin / 5mg dapagliflozin / 1000 mg metformin XR without food.
  Interventions: Drug: 2.5 mg Saxagliptin tablet; Drug: 5 mg dapagliflozin / 1000 mg metformin XR tablet; Drug: Triple FCDP - 2.5 mg saxagliptin / 5 mg dapagliflozin / 1000 mg metformin XR
- Cohort 2: Sequence 1 (DEF) (Experimental): Subjects were randomized to treatment sequence 1 ABC:
  On Day 1, each subjects will receive orally single-dose of the treatment assigned to that treatment period.
  D= Reference product - 5mg ONGLYZA (5mg saxagliptin) and 10/1000mg XIGDUO XR (10 mg dapagliflozin / 1000mg Metformin XR) after food.
  E = Test product - Triple FCDP consisting of 5 mg saxagliptin / 10 mg dapagliflozin / 1000 mg metformin XR after food.
  F = Test product - Triple FCDP tablet consisting of 5 mg saxagliptin / 10 mg dapagliflozin / 1000 mg metformin XR without food.
  Interventions: Drug: 5 mg saxagliptin; Drug: 10 mg dapagliflozin / 1000 mg metformin XR tablet; Drug: Triple FCDP - 5 mg saxagliptin / 10 mg dapagliflozin / 1000 mg metformin XR
- Cohort 2: Sequence 2 (DFE) (Experimental): Subjects were randomized to treatment sequence 1 ABC:
  On Day 1, each subjects will receive orally single-dose of the treatment assigned to that treatment period.
  D= Reference product - 5mg ONGLYZA (5mg saxagliptin) and 10/1000mg XIGDUO XR (10 mg dapagliflozin / 1000mg Metformin XR) after food.
  E = Test product - Triple FCDP consisting of 5 mg saxagliptin / 10 mg dapagliflozin / 1000 mg metformin XR after food.
  F = Test product - Triple FCDP tablet consisting of 5 mg saxagliptin / 10 mg dapagliflozin / 1000 mg metformin XR without food.
  Interventions: Drug: 5 mg saxagliptin; Drug: 10 mg dapagliflozin / 1000 mg metformin XR tablet; Drug: Triple FCDP - 5 mg saxagliptin / 10 mg dapagliflozin / 1000 mg metformin XR
- Cohort 2: Sequence 3 (EDF) (Experimental): Subjects were randomized to treatment sequence 1 ABC:
  On Day 1, each subjects will receive orally single-dose of the treatment assigned to that treatment period.
  D= 5mg ONGLYZA (5mg saxagliptin) and 10/1000mg XIGDUO XR (10 mg dapagliflozin / 1000mg Metformin XR) after food.
  E = Triple FCDP consisting of 5 mg saxagliptin / 10 mg dapagliflozin / 1000 mg metformin XR after food.
  F = Triple FCDP tablet consisting of 5 mg saxagliptin / 10 mg dapagliflozin / 1000 mg metformin XR without food.
  Interventions: Drug: 5 mg saxagliptin; Drug: 10 mg dapagliflozin / 1000 mg metformin XR tablet; Drug: Triple FCDP - 5 mg saxagliptin / 10 mg dapagliflozin / 1000 mg metformin XR
- Cohort 2: Sequence 4 (EFD) (Experimental): Subjects were randomized to treatment sequence 1 ABC:
  On Day 1, each subjects will receive orally single-dose of the treatment assigned to that treatment period.
  D= Reference product - 5mg ONGLYZA (5mg saxagliptin) and 10/1000mg XIGDUO XR (10 mg dapagliflozin / 1000mg Metformin XR) after food.
  E = Test product - Triple FCDP consisting of 5 mg saxagliptin / 10 mg dapagliflozin / 1000 mg metformin XR after food.
  F = Test product - Triple FCDP tablet consisting of 5 mg saxagliptin / 10 mg dapagliflozin / 1000 mg metformin XR without food.
  Interventions: Drug: 5 mg saxagliptin; Drug: 10 mg dapagliflozin / 1000 mg metformin XR tablet; Drug: Triple FCDP - 5 mg saxagliptin / 10 mg dapagliflozin / 1000 mg metformin XR
- Cohort 2: Sequence 5 (FDE) (Experimental): Subjects were randomized to treatment sequence 1 ABC:
  On Day 1, each subjects will receive orally single-dose of the treatment assigned to that treatment period.
  D= Reference product - 5mg ONGLYZA (5mg saxagliptin) and 10/1000mg XIGDUO XR (10 mg dapagliflozin / 1000mg Metformin XR) after food.
  E = Test product - Triple FCDP consisting of 5 mg saxagliptin / 10 mg dapagliflozin / 1000 mg metformin XR after food.
  F = Test product - Triple FCDP tablet consisting of 5 mg saxagliptin / 10 mg dapagliflozin / 1000 mg metformin XR without food.
  Interventions: Drug: 5 mg saxagliptin; Drug: 10 mg dapagliflozin / 1000 mg metformin XR tablet; Drug: Triple FCDP - 5 mg saxagliptin / 10 mg dapagliflozin / 1000 mg metformin XR
- COhort 2: Sequence 6 (FED) (Experimental): Subjects were randomized to treatment sequence 1 ABC:
  On Day 1, each subjects will receive orally single-dose of the treatment assigned to that treatment period.
  D= Reference product - 5mg ONGLYZA (5mg saxagliptin) and 10/1000mg XIGDUO XR (10 mg dapagliflozin / 1000mg Metformin XR) after food.
  E = Test product - Triple FCDP consisting of 5 mg saxagliptin / 10 mg dapagliflozin / 1000 mg metformin XR after food.
  F = Test product - Triple FCDP tablet consisting of 5 mg saxagliptin / 10 mg dapagliflozin / 1000 mg metformin XR without food.
  Interventions: Drug: 5 mg saxagliptin; Drug: 10 mg dapagliflozin / 1000 mg metformin XR tablet; Drug: Triple FCDP - 5 mg saxagliptin / 10 mg dapagliflozin / 1000 mg metformin XR

INTERVENTIONS:
Drug: 2.5 mg Saxagliptin tablet — A competitive dipeptidyl peptidase-4 (DPP-4) inhibitor, slows the inactivation of the incretin hormones, thereby increases their bloodstream concentrations and reduces fasting and post-prandial glucose concentrations in a glucose-dependent manner in subjects with Type 2 diabetes mellitus (T2DM).
  Other Names: 2.5 mg ONGLYZA
  Arms: Cohort 1: Sequence 1 (ABC); Cohort 1: Sequence 2 (ACB); Cohort 1: Sequence 3 (BAC); Cohort 1: Sequence 4 (BCA); Cohort 1: Sequence 5 (CAB); Cohort 1: Sequence 6 (CBA)
Drug: 5 mg dapagliflozin / 1000 mg metformin XR tablet — Dapagliflozin - An inhibitor of sodium-glucose co-transporter 2 (SGLT-2), reduces re-absorption of filtered glucose and lowers the renal threshold for glucose, and thereby increases urinary glucose excretion.
  Metformin - Lowers both basal and post-prandial plasma glucose by decreasing hepatic glucose production and intestinal absorption of glucose; improves insulin sensitivity by increasing peripheral glucose uptake and utilization.
  Other Names: 5 / 1000 mg XIGDUO XR
  Arms: Cohort 1: Sequence 1 (ABC); Cohort 1: Sequence 2 (ACB); Cohort 1: Sequence 3 (BAC); Cohort 1: Sequence 4 (BCA); Cohort 1: Sequence 5 (CAB); Cohort 1: Sequence 6 (CBA)
Drug: Triple FCDP - 2.5 mg saxagliptin / 5 mg dapagliflozin / 1000 mg metformin XR — Saxagliptin - A competitive dipeptidyl peptidase-4 (DPP-4) inhibitor, slows the inactivation of the incretin hormones, thereby increases their bloodstream concentrations and reduces fasting and post-prandial glucose concentrations in a glucose-dependent manner in subjects with T2DM.
  Dapagliflozin - An inhibitor of SGLT-2, reduces re-absorption of filtered glucose and lowers the renal threshold for glucose, and thereby increases urinary glucose excretion.
  Metformin - Lowers both basal and post-prandial plasma glucose by decreasing hepatic glucose production and intestinal absorption of glucose; improves insulin sensitivity by increasing peripheral glucose uptake and utilization.
  Arms: Cohort 1: Sequence 1 (ABC); Cohort 1: Sequence 2 (ACB); Cohort 1: Sequence 3 (BAC); Cohort 1: Sequence 4 (BCA); Cohort 1: Sequence 5 (CAB); Cohort 1: Sequence 6 (CBA)
Drug: 5 mg saxagliptin — A competitive dipeptidyl peptidase-4 (DPP-4) inhibitor, slows the inactivation of the incretin hormones, thereby increases their bloodstream concentrations and reduces fasting and post-prandial glucose concentrations in a glucose-dependent manner in subjects with T2DM.
  Other Names: 5 mg ONGLYZA
  Arms: COhort 2: Sequence 6 (FED); Cohort 2: Sequence 1 (DEF); Cohort 2: Sequence 2 (DFE); Cohort 2: Sequence 3 (EDF); Cohort 2: Sequence 4 (EFD); Cohort 2: Sequence 5 (FDE)
Drug: 10 mg dapagliflozin / 1000 mg metformin XR tablet — Dapagliflozin - An inhibitor of SGLT-2, reduces re-absorption of filtered glucose and lowers the renal threshold for glucose, and thereby increases urinary glucose excretion.
  Metformin - Lowers both basal and post-prandial plasma glucose by decreasing hepatic glucose production and intestinal absorption of glucose; improves insulin sensitivity by increasing peripheral glucose uptake and utilization.
  Other Names: 10/1000 mg XIGDUO XR
  Arms: COhort 2: Sequence 6 (FED); Cohort 2: Sequence 1 (DEF); Cohort 2: Sequence 2 (DFE); Cohort 2: Sequence 3 (EDF); Cohort 2: Sequence 4 (EFD); Cohort 2: Sequence 5 (FDE)
Drug: Triple FCDP - 5 mg saxagliptin / 10 mg dapagliflozin / 1000 mg metformin XR — Saxagliptin - A competitive dipeptidyl peptidase-4 (DPP-4) inhibitor, slows the inactivation of the incretin hormones, thereby increases their bloodstream concentrations and reduces fasting and post-prandial glucose concentrations in a glucose-dependent manner in subjects with T2DM.
  Dapagliflozin - An inhibitor of SGLT-2, reduces re-absorption of filtered glucose and lowers the renal threshold for glucose, and thereby increases urinary glucose excretion.
  Metformin - Lowers both basal and post-prandial plasma glucose by decreasing hepatic glucose production and intestinal absorption of glucose; improves insulin sensitivity by increasing peripheral glucose uptake and utilization.
  Arms: COhort 2: Sequence 6 (FED); Cohort 2: Sequence 1 (DEF); Cohort 2: Sequence 2 (DFE); Cohort 2: Sequence 3 (EDF); Cohort 2: Sequence 4 (EFD); Cohort 2: Sequence 5 (FDE)

SUMMARY:
A Study to Assess the Fed-state Bioequivalence of a Triple Fixed-Combination Drug Product (FCDP) of 2.5 mg Saxagliptin / 5 mg Dapagliflozin / 1000 mg Metformin XR and 5 mg Saxagliptin /10 mg Dapagliflozin /1000 mg Metformin XR Relative to Individual Components (Onglyza and XIGDUO XR) Co-administration. A randomized, open-label, cross over design has been chosen to minimize the effects of between-subject variability and any period effects on the overall results.

DETAILED DESCRIPTION:
This study will be randomized, 3-period, 3-treatment, single-dose, open-label, single-center, crossover to assess the fed-state bioequivalence of a two triple Fixed-combination Drug Product (FCDP) of saxagliptin/dapagliflozin/metformin extended-release (XR) relative to individual components co-administered in approximately 84 healthy adult subjects. Eligible subjects will be healthy male and female aged 18 to 55 years, with a body weight of 50 to 100 kg and body mass index (BMI) of 18 to 32 kg/m2. Of the 84 randomized subjects (2 cohorts of 42 subjects each [3 treatments in each cohort]), at least 72 subjects (36 in each cohort) should be evaluable. Each randomized subject will receive 3 single-dose treatments and each treatment will be administered within 1 of the 3 successive treatment periods. Within each cohort subjects will be randomized to 1 to 6 treatment sequences prescribing the ordered sequence of 3 administered treatments with 7 subjects in each treatment sequence. The investigational medicinal product (IMPs) will be administered orally at single-dose to subjects within 5 minutes after standard meal (light-fat, low-calorie) in the morning (fed condition) or following a 10 hour fast (fasted condition). In both cohorts, test product will be compared with treatments of fed and fasted conditions Subjects in Cohort 1 will be randomized to one of the treatment sequences (ABC), (ACB), (BAC), (BCA), (CAB) or (CBA).

Treatment A (Reference Product under fed conditions) - Single-dose of 2.5 mg saxagliptin (ONGLYZA) and 5 mg dapagliflozin / 1000 mg metformin XR (XIGDUO XR) tablets.

Treatment B (Test Product under fed conditions) - Single-dose of triple FCDP consisting of 2.5 mg saxagliptin / 5 mg dapagliflozin / 1000 mg metformin XR.

Treatment C (Test Product fasted conditions) - Single-dose of triple FCDP tablet consisting of 2.5 mg saxagliptin / 5 mg dapagliflozin / 1000 mg metformin XR.

Subjects in Cohort 2 will be randomized to one of the treatment sequences (DEF), (DFE), (EDF), (EFD), (FDE) or (FED).

Treatment D (Reference product under fed conditions) - Single-dose of 5 mg saxagliptin (ONGLYZA) and 10 mg dapagliflozin / 1000 mg metformin XR (XIGDUO XR) tablet.

Treatment E (Test Product under fed conditions) - Single-dose of triple FCDP consisting of 5 mg saxagliptin / 10 mg dapagliflozin / 1000 mg metformin XR.

Treatment F (Test Product under fasted conditions) - Single-dose of triple FCDP consisting of 5 mg saxagliptin / 10 mg dapagliflozin / 1000 mg metformin XR.

The study will comprise:

* A screening period of maximum 28 days;
* Three resident treatment periods - Day before dosing with the IMP (Day -1) until at least 72 hours after dosing; and will be discharged on the morning of Day 4; and
* A follow-up visit within 5 to 7 days after the last dose of IMP. Treatment periods will be separated by a minimum washout period of 7 to 14 days between each IMP dose. The duration of the study will be approximately 7 to 9 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent prior to any study specific procedures.
2. Healthy male and/or female subjects aged 18 to 55 years with suitable veins for cannulation or repeated venipuncture.
3. Female subject must have a negative serum pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin) at Screening and negative urine pregnancy test within 24 hours prior to investigational medicinal product (IMP) administration and either: a) Be of non-childbearing potential, confirmed at screening by fulfilling one of the following criteria: - Postmenopausal defined as amenorrhea for at least 12 months or more following cessation of all exogenous hormonal treatments and FSH levels in the postmenopausal range.

   - Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation.

   b). Or, if of childbearing potential: - Must not be nursing (breastfeeding). -And, if heterosexually active, agree to consistently use an acceptable method of contraception to avoid pregnancy, from at least 4 weeks prior to dosing and throughout the study and for up to 90 days after the last dose of IMP.
4. Sexually active fertile male subjects must use effective birth control for the entire study and 90 days after the last dose of IMP if their partners are women of childbearing potential.
5. Have a body mass index (BMI) between 18 and 32 kg/m2 inclusive and weigh at least 50 kg and no more than 100 kg inclusive.

Exclusion Criteria:

1. History of any clinically significant disease or disorder which, in the opinion of the principal investigator (PI), may either put the volunteer at risk because of participation in the study, or influence the results or the volunteer's ability to participate in the study.
2. Current or recent (within 3 months of first IMP dosing) gastrointestinal (GI) disease that may impact drug absorption and affect the PK of the study drugs. Additionally, any GI surgery (e.g., partial gastrectomy, pyloroplasty) including cholecystectomy that may impact drug absorption.
3. Any major surgery, as determined by the investigator, within 4 weeks of first IMP dosing.
4. Donation of > 400 mL of blood within 8 weeks or donation of plasma (except at the Screening Visit) within 4 weeks of first IMP dosing.
5. Blood transfusion within 4 weeks of first IMP dosing.
6. Inability to tolerate oral medication.
7. Inability to tolerate venipuncture or inadequate venous access as determined by the investigator.
8. Recent (within 6 months of first IMP dosing) drug or alcohol abuse as defined in the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV), Diagnostic Criteria for Drug and Alcohol Abuse.
9. Subjects who drink more than 3 cups of coffee or other caffeine-containing products a day, or 5 cups of tea a day.
10. Use of tobacco-containing or nicotine-containing products (including but not limited to cigarettes, pipes, cigars, chewing tobacco, nicotine patches, nicotine lozenges, or nicotine gum) within 6 months prior to first check-in (Day -1, Treatment Period 1), or a positive nicotine test (i.e., cotinine) at Screening and/or check-in.
11. History of diabetes mellitus, heart failure, chronic or recurrent urinary tract infection (defined as 3 occurrences per year) and severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the PI or history of hypersensitivity to drugs with a similar chemical structure or class to saxagliptin, dapagliflozin and metformin.

14. Recent vulvovaginal mycotic infection (within 2 months prior to first IMP dosing).

15. Any other sound medical, psychiatric and/or social reason as determined by the investigator.

16. Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of Screening.

17. Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody, and human immunodeficiency virus (HIV) antibody.

18. Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 3 months of the first administration of IMP in this study. The period of exclusion begins 3 months after the final dose or one month after the last visit whichever is the longest.

19. Positive screen for drugs of abuse or cotinine at Screening or on each admission to the clinical unit or positive screen for alcohol on each admission to the clinical unit.

20. Use of saxagliptin, dapagliflozin and/or metformin within 3 months prior to the first administration of IMP.

21. Use of any prescription drugs or over the counter acid controllers within 4 weeks prior to the first administration of IMP except medication cleared by the medical monitor.

22. Use of drugs with enzyme-inducing properties such as St John's Wort within 3 weeks prior to the first administration of IMP.

23. Use of any prescribed or non-prescribed medication including analgesics (other than paracetamol / acetaminophen), herbal remedies, megadose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during the 2 weeks prior to the first administration of IMP or longer if the medication has a long half-life. Note: Hormonal replacement therapy is not allowed.

24. Involvement of any AstraZeneca, PAREXEL or study site employee or their close relatives.

25. Vulnerable subjects, e.g., kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 85 (Actual)
Dates: Start 2017-05-29 (Actual); Primary Completion 2017-08-03 (Actual); Study Completion 2017-08-03 (Actual)

PRIMARY OUTCOMES:
Area under plasma concentration-time curve from time zero to infinity (AUC) | Day 1 to Day 4 (At pre-dose and post-dose at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 18, 24, 36, 48, 60 and 72 hours)
  To assess pharmacokinetics (PK) in terms of AUC in Cohort 1 after administration of Treatment A, B (under fed condition), C (under fasted condition) and Cohort 2 after administration of Treatment D, E (under fed condition) and F (under fasted condition) in healthy volunteers.
Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration (AUC0-t) | Day 1 to Day 4 (At pre-dose and post-dose at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 18, 24, 36, 48, 60 and 72 hours)
  To assess PK in terms of AUC0-t in Cohort 1 after administration of Treatment A, B (under fed condition), C (under fasted condition) and Cohort 2 after administration of Treatment D, E (under fed condition) and F (under fasted condition) in healthy volunteers.
Maximum observed plasma concentration (Cmax) | Day 1 to Day 4 (At pre-dose and post-dose at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 18, 24, 36, 48, 60 and 72 hours)
  To assess PK in terms of Cmax in Cohort 1 after administration of Treatment A, B (under fed condition), C (under fasted condition) and Cohort 2 after administration of Treatment D, E (under fed condition) and F (under fasted condition) in healthy volunteers.

SECONDARY OUTCOMES:
Time to reach maximum observed plasma concentration (tmax) | At pre-dose and post-dose at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 18, 24, 36, 48, 60 and 72 hours
  To assess PK in terms of tmax in Cohort 1 after administration of Treatment A, B (under fed condition), C (under fasted condition) and Cohort 2 after administration of Treatment D, E (under fed condition) and F (under fasted condition) in healthy volunteers.
Half-life associated with terminal slope (λz) of a semi-logarithmic concentration-time curve (t1/2) | At pre-dose and post-dose at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 18, 24, 36, 48, 60 and 72 hours
  To assess PK in terms of t1/2 in Cohort 1 after administration of Treatment A, B (under fed condition), C (under fasted condition) and Cohort 2 after administration of Treatment D, E (under fed condition) and F (under fasted condition) in healthy volunteers.
Mean residence time of the unchanged drug in the systemic circulation from zero to infinity (parent drug only) (MRT) | At pre-dose and post-dose at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 18, 24, 36, 48, 60 and 72 hours
  To assess PK in terms of MRT in Cohort 1 after administration of Treatment A, B (under fed condition), C (under fasted condition) and Cohort 2 after administration of Treatment D, E (under fed condition) and F (under fasted condition) in healthy volunteers.
Terminal elimination rate constant (λz) | At pre-dose and post-dose at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 18, 24, 36, 48, 60 and 72 hours
  To assess PK in terms of λz in Cohort 1 after administration of Treatment A, B (under fed condition), C (under fasted condition) and Cohort 2 after administration of Treatment D, E (under fed condition) and F (under fasted condition) in healthy volunteers.
Apparent total body clearance of drug from plasma after extravascular administration (CL/F) | At pre-dose and post-dose at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 18, 24, 36, 48, 60 and 72 hours
  To assess PK in terms of CL/F in Cohort 1 after administration of Treatment A, B (under fed condition), C (under fasted condition) and Cohort 2 after administration of Treatment D, E (under fed condition) and F (under fasted condition) in healthy volunteers.
Apparent volume of distribution (V/F) | At pre-dose and post-dose at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 18, 24, 36, 48, 60 and 72 hours
  To assess PK in terms of V/F in Cohort 1 after administration of Treatment A, B (under fed condition), C (under fasted condition) and Cohort 2 after administration of Treatment D, E (under fed condition) and F (under fasted condition) in healthy volunteers.
Ratio of metabolite AUC to parent AUC (MRAUC) | At pre-dose and post-dose at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 18, 24, 36, 48, 60 and 72 hours
  To assess PK in terms of MRAUC in Cohort 1 after administration of Treatment A, B (under fed condition), C (under fasted condition) and Cohort 2 after administration of Treatment D, E (under fed condition) and F (under fasted condition) in healthy volunteers.
Number of subjects with Adverse Events (AEs) | A Day -1, spontaneous plus pre-dose, 1, 2, 3, 24, and 48 hours post-dose
  To assess AEs as a criteria of safety and tolerability variables.
Systolic and diastolic blood pressure [BP] | At screening (Day -28), Day -1, pre-dose, 71 hours post-dose and 5 to 7 days post-final dose follow-up
  To assess the systolic and diastolic blood pressure as a criteria of safety and tolerability variables
Pulse rate | From Screening (Day -28 to Day -1) to Follow-up (5-7days post final dose)
  To assess the pulse rate as a criteria of safety and tolerability variables
Twelve-lead electrocardiograms (ECGs) | From Screening (Day -28 to Day -1) to Follow-up (5-7days post final dose)
  To assess the cardiovascular system functioning as a criteria of safety and tolerability variables.
Physical examination | From Screening (Day -28 to Day -1) to Follow-up (5-7days post final dose)
  To assess a complete physical examinations (general appearance, respiratory, cardiovascular, abdomen, skin, head, and neck (including ears, eyes, nose and throat), lymph nodes, thyroid, musculoskeletal and neurological systems) and a brief physical examinations (general appearance, skin, abdomen, cardiovascular system and respiratory) as a criteria of safety and tolerability variables.
  A complete physical examination will be performed at the screening visit.
Laboratory assessments of Hematology | From Screening (Day -28 to Day -1) to Follow-up (5-7days post final dose)
  To assess the count of white blood cell (WBC), red blood cell (RBC) and platelets; absolute count of neutrophils, lymphocytes, monocytes, eosinophils, basophils and reticulocytes; levels of Hemoglobin (Hb), hematocrit (HCT), mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH) and mean corpuscular hemoglobin concentration (MCHC) in blood as a criteria of safety and tolerability variables.
Laboratory assessments of Clinical chemistry | From Screening (Day -28 to Day -1) to Follow-up (5-7days post final dose)
  To assess the levels of electrolytes (sodium, potassium, magnesium, chloride, calcium, phosphate), urea, creatinine, albumin, glucose (fasting), C-reactive protein (CRP), thyroxine (T4), thyroid-stimulating hormone (TSH), liver enzymes (alkaline phosphatase (ALP), alanine aminotransferase (ALT), aspartate aminotransferase (AST) and Gamma glutamyl transpeptidase (GGT)), bilirubin (total and unconjugated) and follicle-stimualting hormone (FSH) in serum as a criteria of safety and tolerability variables.
Laboratory assessments of urinalysis | From Screening (Day -28 to Day -1) to Follow-up (5-7days post final dose)
  To assess the presence of glucose, protein, blood and microscopy (RBC, WBC, casts (cellualr, granular, hyaline) in urine as a criteria of safety and tolerability variables.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Tang W, Engman H, Zhu Y, Dayton B, Boulton DW. Bioequivalence and Food Effect of Dapagliflozin/Saxagliptin/Metformin Extended-release Fixed-combination Drug Products Compared With Coadministration of the Individual Components in Healthy Subjects. Clin Ther. 2019 Aug;41(8):1545-1563. doi: 10.1016/j.clinthera.2019.05.015. Epub 2019 Jun 29. PMID 31266654